CLINICAL TRIAL: NCT03561974
Title: Impact of Humidification on Sleep Quality During Home Non Invasive Ventilation
Acronym: IMHUNIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMHUNIV
Record Dates: First submitted 2018-05-18; First posted 2018-06-19 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Chronic Respiratory Failure With Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Humidification (Experimental)
  Interventions: Device: Humidification
- Control group without humidification (No Intervention)

INTERVENTIONS:
Device: Humidification — Patients will benefit of humidification and warming of delivered gaz by non-invasive ventilation thanks humidification system.
  Arms: Humidification

SUMMARY:
Protocol Summary:

1. Question Does the adjunction of a humidification system to non-invasive ventilation circuit improve sleep quality and comfort of chronic ventilated respiratory insufficient patients? Does it change the efficacy of long-term non invasive ventilation therapy and patient-ventilator interactions?
2. Aims

Main aim:

The primary endpoint of this study is to objectively evaluate the consequences of a humidification system's adjunction on quality of sleep, 2 months after treatment's beginning.

Second aims:

The secondary endpoints are to evaluate the consequences of a humidification system's adjunction on non invasive ventilation's efficacy / patient-ventilator asynchronies / patients' comfort / treatment adherence.

Before the clinical trial, the investigators conducted a bench study using a mechanical lung in order to evaluate the ventilator's behavior with and without a humidification system.

The clinical trial will include patients with chronic respiratory failure with an indication of long-term non invasive ventilation therapy. Patients will be included in the Pulmonology, Thoracic Oncology and Respiratory intensive care unit of Rouen University Hospital.

It will be a prospective monocentric study, including consecutively all eligible patients. Informed consent will be obtained from all of them.

At baseline, patients will be hospitalized for two consecutive nights for non invasive ventilation's set up. During the first night, a polysomnography will be performed without non invasive ventilation. Then, patients will be treated by non invasive ventilation with a bi-level self-regulated pressure mode and an open circuit.

Patients will be randomized in two groups: without a humidification system and with a humidification system. Partitioning by the physiopathological pattern (obstructive versus obesity hypoventilation syndrome vs. neuromuscular disease) will be done.

During each night, arterial blood gases will be measured at bedtime and awakening. Patients will be monitored by:

* polysomnography (only during the first night)
* transcutaneous capnography
* accessory inspiratory muscles surface electromyography
* pneumotachograph on non invasive ventilation's circuit
* pressions measured at the mask.

Follow-up will take place at two months after non invasive ventilation's beginning with or without humidification. Patients will be hospitalized for one night only. Blood gases at bedtime and at awakening will be measured. A polysomnography with non invasive ventilation will be performed. Observance will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 chronic respiratory failure (PaCO2 > 6,5 at the time of the diagnosis)
* Indication of a long term non invasive ventilation at home because of an obstructive respiratory disease, a obesity hypoventilation syndrome or a neuromuscular disease.
* Over eighteen years old
* Planned hospitalisation to introduce non invasive ventilation.

Exclusion Criteria:

* Less than eighteen years old
* Pregnancy
* Psychiatric or cognitive disorders in wich consent is not possible
* Acute respiratory failure within 2 weeks before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sleep quality at two month | Assessement will be performed at baseline and 2 month after initiation of non invasive ventilation with or without humidification.
  Sleep quality will be assessed by polysomnography without non invasive ventilation at Baseline versus with non invasive ventilation at follow up with or without humification (after 2month)

SECONDARY OUTCOMES:
Subjective sleep quality | Assessement will be performed at baseline and 2 month after initiation of non invasive ventilation with or without humidification.
  Outcome will be assessed using the Pittsburgh sleep quality index. The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a one-month time interval. The measure consists of nineteen individual items, creating seven components which are summed to produce a global score. Each component ranges from zero to three (zero: no difficulty at all ; three: great difficulties). Global score ranges from zero (no difficulty) to twenty-one points (great difficulties).
Nature of patient-ventilator asynchrony | Assessement will be performed at baseline and 2 month after initiation of non invasive ventilation with or without humidification.
  Outcome will be assessed by two independent investigators through raw data from the ventilator
Number of patient-ventilator asynchrony | Assessement will be performed at baseline and 2 month after initiation of non invasive ventilation with or without humidification.
  Outcome will be assessed by two independent investigators through raw data from the ventilator
Comfort with non invasive ventilation | Assessement will be performed at baseline and 2 month after initiation of non invasive ventilation with or without humidification.
  Outcome will be assessed using a visual analogic scale ranging from zero to ten (zero: very uncomfortable ; ten: greater comfort).
Nasal obstruction | Assessement will be performed at baseline and 2 month after initiation of non invasive ventilation with or without humidification.
  Outcome will be assessed using the Nasal Obstruction Symptom Evaluation questionary (NOSE) which is an instrument allowing clinicians to better understand impact of nasal obstruction on patients' quality of life. The measure consists of five individual items evaluated on a one-month past interval. Each item ranges from zero (not a problem) to four (severe problem). Then, scores are summed to create a global score ranging from zero (not a problem) to twenty (severe problem).
Rhinorrhea and xerostomia | Assessement will be performed at baseline and 2 month after initiation of non invasive ventilation with or without humidification.
  Outcomes will be assessed using visual analogic scale ranging from zero to ten (zero: no rhinorrhea or xerostomia at all ; ten: worse rhinorrhea or xerostomia).
Quality of life: Severe Inspirator Insufficiency questionary | Assessement will be performed at baseline and 2 month after initiation of non invasive ventilation with or without humidification.
  Outcome will be assessed using the Severe Inspirator Insufficiency questionary. It's a specific instrument for measuring health-related quality of life in patients receiving home mechanical ventilation. The measure consists of forty-nine individual items, creating seven components which are summed to produce a global score. Each item ranges from one to five (one: not true ; five: very true). Each component ranges from zero to one hundred. Global score is the seven components' mean. It ranges from zero (bad quality of life) to one hundred percent (best quality of life).
Number of nightime disruption of non invasive ventilation | Assessement will be performed at baseline and 2 month after initiation of non invasive ventilation with or without humidification.
  Outcome will be assessed using raw data from the ventilator.
Adherence | Outcome will be assessed at study completion (two months follow-up).
  Number of hours of treatment by night

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Cuvelier, Prof, PhD, Principal Investigator — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France; Maxime Patout, MD, MsC, Principal Investigator — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France; Astrid Bertier, MD, Principal Investigator — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France
Locations (1):
- ADIR Association, Bois-Guillaume, France